CLINICAL TRIAL: NCT00887562
Title: A Phase IIa Double-Blind, Randomized, Placebo-Controlled, Dose-Finding Study of Idebenone in the Treatment of Mitochondrial Encephalopathy Lactic Acidosis and Stroke-like Episodes
Brief Title: Study of Idebenone in the Treatment of Mitochondrial Encephalopathy Lactic Acidosis & Stroke-like Episodes
Acronym: MELAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michio Hirano (Other)
Collaborators: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Michio Hirano, Professor of Neurology, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAC9240; SNT-II-007 (Other: Santhera)
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2016-08-10 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-09

CONDITIONS: MELAS Syndrome
MeSH Terms: conditions — MELAS Syndrome | interventions — idebenone; Bulk Drugs

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Idebenone 900 mg/day (Experimental): Idebenone 900 mg/day
  Interventions: Drug: Idebenone
- Idebenone 2250 mg/day (Experimental): Idebenone 2250 mg/day
  Interventions: Drug: Idebenone
- placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Idebenone — 900 mg/day for 1 month
  Other Names: active drug
  Arms: Idebenone 900 mg/day
Drug: Idebenone — 2250 mg/day for 1 month
  Other Names: active drug
  Arms: Idebenone 2250 mg/day
Other: Placebo — Placebo - No idebenone
  Other Names: No active drug
  Arms: placebo

SUMMARY:
The purpose of this study is to compare the efficacy of two (2) different doses of idebenone with that of a placebo over a one month period on cerebral lactate concentration as measured by magnetic resonance spectroscopy.

DETAILED DESCRIPTION:
MELAS (Mitochondrial Encephalomyopathy, Lactic Acidosis, and Stroke-Like Episodes), a progressive and often devastating multisystem disorder, is most commonly associated with mitochondrial Deoxyribonucleic acid (mtDNA) point mutation at nucleotide 3243. Seizures, cognitive deterioration, and neurobehavioral abnormalities are frequent features of this disease which typically shortens life expectancy. Idebenone, an ATP production modulator and antioxidant, improves neurological function in Friedreich's ataxia, a disease also associated with mitochondrial dysfunction.

Given that there is no effective treatment for MELAS, the investigators propose a Phase II proof of concept trial of idebenone to study its preliminary efficacy in patients with MELAS and the A3243G mtDNA mutation, and to study its safety and tolerability in this patient group.

The investigators propose to evaluate 21 patients with the A3243G mitochondrial DNA mutation and MELAS (defined by a history of either seizures or stroke). Patients will receive idebenone (900 mg/day or 2250 mg/day) or matching placebo for one month. The primary outcome measure is cerebral lactate levels measured by Magnetic Resonance Spectroscopy (MRS), a biomarker associated with disease worsening. This study will help the investigators to determine if there is sufficient signal to proceed to efficacy studies. Also it will provide additional information on the safety and tolerability of two different doses of idebenone in MELAS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MELAS with confirmed A3243G mtDNA mutation, or evidence of central nervous system involvement (cognitive problems, migraines, memory loss)
* Cerebral lactate level equal to or greater than 5.0 i.u. at baseline
* Patients at least 8 and < 65 years of age at baseline
* Patients with a body weight > 37 kg/82 lbs at baseline
* Stable co-medication/vitamins/supplements within 1 month prior to baseline
* Patients who in the opinion of the investigator are able to comply with the requirements of the study, including swallowing the study medication
* Negative urine pregnancy test at screening and baseline (female patients of childbearing potential)

Exclusion Criteria:

* Contraindication to MRS (e.g. metal implant, claustrophobia)
* Stroke like event within 2 months prior to baseline
* Treatment with idebenone at any dose, or coenzyme Q10 at doses above 100mg/d within 1 month prior to baseline
* Inadequate contraception use
* Pregnancy and/or breast-feeding
* Clinically significant abnormalities of clinical hematology or biochemistry including, but not limited to, elevations greater than 1.5 times the upper limit of normal of aspartate aminotransferase (AST), alanine aminotransferase (ALT) or creatinine
* Current abuse of drugs or alcohol
* Participation in a trial of another investigational drug within the last month
* Other factor that, in the investigator's opinion, excludes the patient from entering the study

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michio Hirano, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Idebenone 2250 mg/Day: Idebenone 2250 mg/day
  Idebenone: 2250 mg/day for one month
Period: Overall Study
Arm/Group | Idebenone 900 mg/Day | Idebenone 2250 mg/Day | Placebo
Started | 10 | 9 | 8
Completed | 7 | 7 | 7
Not Completed | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Idebenone 900 mg/Day | Idebenone 2250 mg/Day | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 8 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 1
  Between 18 and 65 years | 9 | 9 | 8 | 26
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 6 | 20
  Male | 1 | 4 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 0 | 3
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 8 | 8 | 23
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 8 | 27

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Cerebral Lactate Concentration (as Measured by Magnetic Resonance Spectroscopy)
Description: To compare the efficacy of 1 month treatment with 2 different doses of idebenone with that of placebo on cerebral lactate concentration as measured by magnetic resonance spectroscopy (MRS)
Time Frame: Up to 4 weeks from baseline
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Idebenone 900 mg/Day | Idebenone 2250 mg/Day | Placebo
Number analyzed (Participants) | 7 | 7 | 7
IU | -0.09 (0.95) | 0.16 (1.49) | -0.49 (1.18)

2. Secondary Outcome: Mean Change in Venous Lactate Concentration
Description: To compare the efficacy of 1 month treatment with 2 different doses of idebenone with that of placebo on venous lactate concentration
Time Frame: Up to 4 weeks from baseline
Measure: Mean (Standard Deviation); unit: mM/L
Arm/Group | Idebenone 900 mg/Day | Idebenone 2250 mg/Day | Placebo
Number analyzed (Participants) | 7 | 7 | 7
mM/L | -0.24 (1.18) | 0.7 (1.31) | -0.46 (1.07)

3. Secondary Outcome: Mean Change in Score on the Fatigue Severity Scale (FSS)
Description: To assess changes following 1 month treatment with 2 different doses of idebenone with that of placebo in fatigue as assessed by the Fatigue Severity Scale (FSS).
  Scale score minimum is 9 (least fatigue) and maximum is 63 (maximum fatigue). Scores of 36 or less indicate possibility that patient may not be suffering from fatigue, while scores 36 and over suggest suffering from fatigue
Time Frame: Baseline and Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 900 mg/Day: Idebenone 900 mg/day
  Idebenone: 900 mg/day for 1 month
- 2250 mg/Day: Idebenone 2250 mg/day
  Idebenone: 2250 mg/day for one month
Arm/Group | 900 mg/Day | 2250 mg/Day | Placebo
Number analyzed (Participants) | 7 | 7 | 7
units on a scale | -3.8 (11) | -1.3 (10) | 4.3 (4.5)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Idebenone 900 mg/Day | Idebenone 2250 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 10/10 | 9/9 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idebenone 900 mg/Day (N=10) | Idebenone 2250 mg/Day (N=9) | Placebo (N=8)
abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
abdominal distention (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (2)
abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (5) | 1 (1)
dispepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
nausea (Gastrointestinal disorders) | 3 (5) | 0 (0) | 0 (0)
chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
fatigue (General disorders) | 5 (8) | 1 (2) | 3 (3)
feeling abnormal (General disorders) | 1 (1) | 1 (1) | 1 (1)
irratibility (General disorders) | 0 (0) | 0 (0) | 1 (2)
lymphadenopathy (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0)
visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (3)
influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
sinusitus (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
albumin in urine (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
bilirubin decreased (Blood and lymphatic system disorders) | 2 (2) | 1 (2) | 1 (1)
chloride decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
creatine phosphokinase increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
glucose decreased (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0)
glucose increase (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
lactic acid increase (Blood and lymphatic system disorders) | 3 (4) | 2 (2) | 2 (2)
carbon dioxide decrease (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 2 (2)
EKG abnormal (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
glucose in urine increased (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
hematocrit decrease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
hemoglobin decrease (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
high density lipoprotein decrease (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
monocyte increased (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
red blood cell decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
ketone in urine increased (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
urine leukocyte esterase increase (Renal and urinary disorders) | 4 (4) | 1 (1) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 1 (2)
headache (Nervous system disorders) | 3 (6) | 2 (2) | 4 (14)
hypoaesthesia (Nervous system disorders) | 1 (2) | 1 (2) | 0 (0)
migraine (Nervous system disorders) | 3 (3) | 0 (0) | 3 (7)
petit mal eplipsey (Nervous system disorders) | 2 (6) | 0 (0) | 1 (1)
somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
nervousness (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1)
pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
lymphadenopathy (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Clinical variability in severity of disease among participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less